CLINICAL TRIAL: NCT02065219
Title: Trigger-point Blockade in Persistent Pain After Open Groin Hernia Repair
Acronym: Trigger-open
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, mads u werner, MD, MDSc, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-3-2011-130-open; 2612-1006 (Other: Danish Medicines Agency)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Inguinal Hernia; Chronic Pain
Keywords: Chronic Pain; Inguinal Hernia; Outcome; Surgical Procedure, Operative
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Experimental): injection, 25 mg, once, 5 min
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): injection, 10 ml 0.9% sodium chloride, once, 5 min
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine — 10 ml of bupivacaine 2.5 mg/ml deposited by ultra-sound guidance around the spermatic cord
  Other Names: Bupivacain "SAD"
  Arms: Bupivacaine
Drug: Placebo — 10 ml 0.9% physiological saline deposited by ultra-sound guidance around the spermatic cord
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Groin hernia repair is a common procedure performed in approximately 2,000 patients per one million inhabitants. Severe chronic pain following groin hernia repair is seen in 2-5% of the patients indicating that a large number of patients each year suffer from debilitating reduction in health-related quality of life.

This study examines the effect of ultra-sound guided blocks with local anesthesia in the groin in regard to pain relief and sleep quality.

The hypothesis of the study is that a block will confer significant pain relief to patients with severe chronic pain following open groin hernia repair.

DETAILED DESCRIPTION:
This placebo-controlled, randomized, double-blind, cross-over study in subjects with severe pain after open groin hernia, examines the effect of an ultra-sound guided local anesthetic block of a trigger-point, situated near the spermatic cord at the superficial inguinal ring. In order to compare effects and distribution of the blocks in patients vs. healthy subjects, the block is tested and examined in volunteers using a similar methodology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent pain (< 6 mo) after open groin hernia repair
* Patients with maximal pain area 3 cm or less from the superficial inguinal ring
* Patients living in the Capital Region of Denmark (Region Hovedstaden) or the Region of Zealand (Region Sjælland)

Exclusion Criteria:

* Known allergy to bupivacaine or other local anesthetics of amide-type
* Declared incapable of making his/hers own affairs
* Does not comprehend Danish in the written or spoken language
* Cognitive impairment to a degree influencing the testing reliability
* Known recurrence of the inguinal hernia
* Other surgical procedures performed in the groin or on the external genitals
* Neuropathy affecting the groin region caused by other conditions, e.g. post-stroke, multiple sclerosis, herniated intervertebral disc
* Abuse of alcohol or drugs
* Unable to cooperate with the sensory examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Normalized summed pain intensity difference (SPID) | 20 min
  The number of patients with normalized summed pain intensity differences (SPID) of more or equal to 50% after bupivacaine AND SPID less or equal to 25% after placebo.

SECONDARY OUTCOMES:
Thermal thresholds | 20 min
  Quantitative changes in thermal thresholds (warmth detection threshold, cool detection thresholds, heat pain threshold) after bupivacaine compared to placebo
Suprathreshold heat stimulation | 20 min
  Quantitative changes in pain ratings to suprathreshold heat stimulation after bupivacaine compared to placebo
Pressure pain thresholds | 20 min
  Quantitative changes in pain rating to pressure algometry stimulation after bupivacaine compared to placebo
Sensory mapping | 20 min
  Quantitative changes in area of cool hypoesthesia assessed by a thermal roller after bupivacaine compared to placebo
Pain questionnaire | 7 days
  Quantitative changes in summed pain intensity differences (SPIDs) during rest, movement and during auto-palpation, assessed morning and evening after bupivacaine compared to placebo
Sleep quality | 7 days
  Quantitative changes in sleep quality assessed each morning, after bupivacaine compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, Principal Investigator — Multidisciplinary Pain Center, Neuroscience Center, Rigshospitalet, Copenhagen University Hospital, DENMARK; Henrik Kehlet, MD, Study Director — Section of Surgical Pathophysiology, Juliane Marie Center, Copenhagen University Hospital, DENMARK
Locations (1):
- Multidisciplinary Pain Center, Neuroscience Center, Copenhagen University Hospital, DENMARK, Copenhagen, Denmark

REFERENCES:
- [Result] Wijayasinghe N, Ringsted TK, Bischoff JM, Kehlet H, Werner MU. The role of peripheral afferents in persistent inguinal postherniorrhaphy pain: a randomized, double-blind, placebo-controlled, crossover trial of ultrasound-guided tender point blockade. Br J Anaesth. 2016 Jun;116(6):829-37. doi: 10.1093/bja/aew071. PMID 27199314